CLINICAL TRIAL: NCT05787574
Title: Phase 2 Study BRIDGING PRE-TRANSPLANT INFLAMMATORY DAMPENING for PRIMARY IMMUNE REGULATORY DISORDERS (BRIDGE Trial)
Brief Title: A Study of Treatment of Inflammation Before Stem Cell Transplant in People With a Primary Immune Regulatory Disorder (PIRD) and/or an Autoinflammatory Condition
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-040; R01FD007829 (FDA)
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Primary Immune Regulatory Disorder; Autoimmune Lymphoproliferative; Immune System Diseases
Keywords: Stem Cell Transplant; Emapalumab; Fludarabine; Dexamethasone; 23-040
MeSH Terms: conditions — Immune System Diseases | interventions — Emapalumab; fludarabine; Dexamethasone; Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: This is a two-stage phase 2 study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Emapalumab (for isolated Interferongamma mediated disease) (Experimental): Participants in this group will receive emapalumab on Days -22 (22 days before the day of the stem cell transplant), -15, -8, and -1.
  Interventions: Drug: Emapalumab; Procedure: Stem Cell Transplant
- Group B: Fludarabine and Dexamethasone (for generalized autoinflammation) (Experimental): Participants in this group will receive fludarabine and dexamethasone for 5 days in a row on Days -22 through -18.
  Interventions: Drug: Fludarabine and Dexamethasone; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Emapalumab — Emapalumab on Days -22 (22 days before the day of the stem cell transplant), -15, -8, and -1.
  Arms: Group A: Emapalumab (for isolated Interferongamma mediated disease)
Drug: Fludarabine and Dexamethasone — Fludarabine and dexamethasone for 5 days in a row on Days -22 through -18.
  Arms: Group B: Fludarabine and Dexamethasone (for generalized autoinflammation)
Procedure: Stem Cell Transplant — Participants in both groups will receive their standard-of-care stem cell transplant on Day 0.

SUMMARY:
The researchers are doing this study to find out whether emapalumab or a combination of fludarabine and dexamethasone are effective in preparing people with a primary immune regulatory disorder (PIRD) and/or an autoinflammatory condition to receive a stem cell transplant. The researchers will look at how well the study treatments reduce inflammation and aid in the engraftment process (the process of donated stem cells traveling to the bone marrow, where they begin to make new immune cells.

"Funding Source - FDA OOPD"

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving first allo-HCT for the following immunologic conditions:
* Primary Immune Regulatory Disorder with or without a genetic lesion as defined by the Primary Immune Deficiency Treatment Consortium (PIDTC)
* Patients with autoinflammatory disorders evidenced by cytokine or inflammation assays with at least 1.5x ULN of measured cytokines and/or an elevated ferritin or ESR > 2 ULN
* For inclusion on the emapalumab group, the lesion must be isolated to the IFNγ pathway (or mediators thereof) with an elevated CXCL9 >1.5 ULN OR sIL2R >1.5 ULN (or already controlled on immune modulation, provided that CXCL9 or sIL2R levels were elevated prior to initiation of immune modulation). Inclusion on the Fludarabine/dexamethasone group requires inflammation (as defined above) other than an isolated IFNγ pathway
* Able to tolerate cytoreduction (based on adequate organ function as described below)
* Patients of any age can enroll so long as they meet other inclusion criteria:
* Adequate organ function is required, defined as follows:

  * Hepatic: Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia. Patients with hyperbilirubinemia related to paroxysmal nocturnal hemoglobinuria or other hemolytic disorders related to their PIRD diagnosis are eligible.
  * Hepatic: AST, ALT, and alkaline phosphatase < 2.5 times the upper limit of normal unless thought to be disease-related. Investigator will need to perform clinically indicated evaluations to assess if disease related or intrinsic liver disease. Additional testing may be done if clinically indicated, after the pre-transplant immune prophase and prior to start of conditioning as this will provide additional data to confirm disease related versus intrinsic liver dysfunction.
  * Renal: serum creatinine <1.5x normal for age. If serum creatinine is outside the normal range, then CrCl > 50 mL/min/1.73m2 (calculated or estimated) or GFR (mL/min/1.72m2) >30% of predicted normal for age.
  * Normal GFR by Age
  * Cardiac: LVEF ≥ 50% by MUGA or resting echocardiogram.
  * Pulmonary: Pulmonary function testing (FEV1 and corrected DLCO) ≥ 50% predicted (pediatric patients unable to complete PFTs will need oxygen saturation as recorded by pulse oximetry of ≥92% on room air).
* Adequate performance status:

  * Age ≥ 16 years: ECOG ≤ 1 or Karnofsky 70%
  * Age < 16 years: Lansky 70%
* Each patient must be willing to participate as a research subject and must sign an informed consent form or legal guardian with assent as appropriate.

Exclusion Criteria:

* Uncontrolled infection at the time of enrollment.
* Patients who have undergone previous allo-HCT.
* Patient seropositivity for HIV I/II and/or HTLV I/II.
* Females who are pregnant or breastfeeding.
* Patients unwilling to use contraception during the study period.
* Patient or parent or guardian unable to give informed consent or unable to comply with the treatment protocol including research tests.

Donor Inclusion Criteria:

* Related Donors:

  * 8/8 or 7/8 HLA matched at A, B, C, and DRB1 loci, as tested by DNA analysis.
  * Haploidentical donors at A, B, C and DRB1 loci, as tested by DNA analysis
* Unrelated Donors:

  o 8/8 or 7/8 matched at A, B, C, and DRB1 loci, as tested by DNA analysis.
* Able to provide informed consent for the donation process per institutional standards.
* Meet standard criteria for donor collection (e.g. National Marrow Donor Program Guidelines or collecting center guidelines as approved by treating physician).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Engraftment | 1 year
  is defined as the first of three days of absolute neutrophil count >500k/µL and the first of seven days of platelets >20,000/µL in the absence of transfusional support.

SECONDARY OUTCOMES:
Determine Overall Survival (OS) | 5 years
  the duration of time between HCT and death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andromachi Scaradavou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - University of California, San Francisco (Data collection only), San Francisco, California
  - Children's Healthcare of Atlanta (Data Collection Only), Atlanta, Georgia
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York
  - Children's Hospital of Philadelphia (Data Collection Only), Philadelphia, Pennsylvania
  - Texas Children's Hospital (Data Collection), Houston, Texas
  - Children's Hospital of Wisconsin (Data Collection Only), Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm